CLINICAL TRIAL: NCT07200661
Title: The Effects of Transcranial Direct Current Stimulation on Improving Impairment and Functional Activity in Individuals With Stroke: A Randomized Controlled Trial
Brief Title: Transcranial Direct Current Stimulation, Functional Activity, Stroke, RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Phayao (Other)
Responsible Party: Principal Investigator, Chonticha Kaewjoho, Lecturer, Department of Physical Therapy, University of Phayao
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UPhayaoChonticha-219
Record Dates: First submitted 2025-09-11; First posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Ischemic Stroke; Hemorrhagic Stroke; Stroke, Cardiovascular
Keywords: Stroke; tDCS; Dual task training; Unstable surfaces; Cognitive function
MeSH Terms: conditions — Ischemic Stroke; Hemorrhagic Stroke; Myocardial Infarction; Stroke

STUDY DESIGN:
Intervention Model Description: Participants will be randomized into three groups. Group A will receive active anodal tDCS (2 mA, 20 min) combined with dual-task stepping on unstable surfaces and overground walking with backward counting. Group B will perform the same dual-task stepping and walking but receive sham tDCS (device switched off after initial ramp-up). Group C will receive active anodal tDCS alone with no motor or cognitive tasks. Interventions will be conducted three times per week for four weeks, totaling 12 sessions. This design allows comparison of combined stimulation and training, training with sham stimulation, and stimulation alone to determine their relative effects on functional ability, walking speed, endurance, lower limb strength, and cognitive outcomes in stroke survivors.
  Intervention frequency: 3 sessions per week (Before and after each exercise session, volunteers' vital signs (blood pressure, oxygen saturation, heart rate) were measured.)
  Program length: 4 weeks
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dual talk with overground walking training + Unstable surface + tDCS (Experimental): Dual talk with overground walking training + Unstable surface + tDCS Volunteers received 10 min of unstable stepping training and 10 min of dual task overground walking training. After that, they received 20 min of transcranial direct current stimulation.
  Note; tDCS: Transcranial direct current stimulation.
  Interventions: Device: Experimental A tDCS: Transcranial direct current stimulation.
- Dual talk with overground walking training + Unstable surface + tDCS (sham) (Sham Comparator): Volunteers received 10 min of unstable stepping training and 10 min of dual task overground walking training. After that, subjects were placed on the head with no electrical current applied for 20 min.
  Note; tDCS: Transcranial direct current stimulation.
  Interventions: Device: Experimental B tDCS: Transcranial direct current stimulation.
- tDCS only (Experimental): Participants in this group will receive anodal tDCS only, without any dual-task or stepping training.
  Electrode placement and stimulation parameters are identical to Group 1 (anodal over ipsilesional M1, reference over contralesional supraorbital area, 2 mA, 20 minutes, with ramp-up and ramp-down). During stimulation, participants will remain seated and relaxed without additional motor or cognitive tasks.
  Total session duration: 20 minutes.
  Interventions: Device: Experimental C tDCS: Transcranial direct current stimulation.

INTERVENTIONS:
Device: Experimental A tDCS: Transcranial direct current stimulation. — Group 1: Active tDCS combined with dual-task stepping (Experimental A) Participants in this group will receive anodal tDCS applied over the ipsilesional primary motor cortex (M1) at C3 or C4 (based on the 10-20 EEG system), with the reference electrode positioned over the contralesional supraorbital area. Stimulation will be delivered at an intensity of 2 mA for 20 minutes, During the stimulation period, participants will perform dual-task stepping exercises on unstable surfaces. The stepping program stepping on a foam pad (5 cm thick, 20 cm wide, 12 cm long). Each stepping session lasts 10 minutes and is immediately followed by overground walking at a comfortable speed for 10 meters, while simultaneously performing a cognitive task of counting backwards from 99 to 0. Participants are instructed not to pause or stop while performing the dual task. If they stop for more than 5 seconds, it is considered an error, which will be recorded.
  Other Names: Unstable surface
  Arms: Dual talk with overground walking training + Unstable surface + tDCS
Device: Experimental B tDCS: Transcranial direct current stimulation. — Group 2:This group follows the same stepping and dual-task walking program as Group 1 (stepping on foam pad for 10 minutes, followed by overground walking with backward counting for 10 minutes). However, instead of active stimulation, participants receive sham tDCS.
  Other Names: Sham tDCS; Unstable surface
  Arms: Dual talk with overground walking training + Unstable surface + tDCS (sham)
Device: Experimental C tDCS: Transcranial direct current stimulation. — Group 3:Participants in this group will receive anodal tDCS only, without any dual-task or stepping training.
  Arms: tDCS only

SUMMARY:
Stroke patients often experience impaired balance and weight-bearing due to muscle weakness and neurological deficits. Motor rehabilitation is a crucial goal in their recovery, and transcranial direct current stimulation (tDCS) has emerged as a promising therapeutic approach. When combined with motor training, tDCS can enhance walking and balance abilities. However, there is a lack of research exploring the combination of unstable surfaces training, cognitive function, and tDCS for stroke rehabilitation

DETAILED DESCRIPTION:
Stroke is a leading cause of long-term disability worldwide, often resulting in impaired motor function, reduced walking ability, decreased muscle strength, and cognitive deficits. These limitations contribute to difficulties in activities of daily living, impaired balance, and reduced quality of life. Effective rehabilitation strategies are essential to promote functional recovery and reduce the risk of long-term dependence.

Transcranial direct current stimulation (tDCS) has emerged as a promising non-invasive neuromodulation technique to facilitate cortical excitability and enhance neuroplasticity in individuals with stroke. Anodal stimulation over the lesioned hemisphere has been shown to improve motor performance and cognitive processing, while sham stimulation does not induce comparable effects. Recent studies suggest that combining tDCS with task-specific rehabilitation programs may provide synergistic benefits by simultaneously enhancing neural activation and functional task performance.

Dual-task training, particularly stepping exercises performed on unstable surfaces, has been demonstrated to challenge both motor and cognitive systems simultaneously. This approach targets balance, gait adaptation, and executive function by requiring patients to divide attention between locomotion and cognitive demands. When applied in combination with tDCS, dual-task training may enhance neuroplasticity and strengthen functional outcomes beyond those achieved by conventional training alone.

The present randomized controlled trial is designed to investigate the combined effects of anodal tDCS and dual-task stepping exercise on unstable surfaces in stroke survivors. Participants will be randomized into three groups: (1) active tDCS combined with dual-task stepping, (2) dual-task stepping with sham tDCS, and (3) active tDCS alone. Interventions will be delivered three times per week for four weeks.

Primary outcomes will include measures of functional ability, walking speed, walking endurance, lower limb muscle strength, and cognitive ability. Secondary outcomes will explore the effects of combined stimulation on balance and overall motor recovery. It is hypothesized that participants receiving combined anodal tDCS and dual-task training will demonstrate greater improvements in both motor and cognitive outcomes compared with either intervention alone.

This study will contribute novel evidence to stroke rehabilitation research by addressing the knowledge gap regarding the integration of non-invasive brain stimulation with cognitive-motor dual-task training on unstable surfaces. The findings are expected to provide insights into effective multimodal rehabilitation strategies aimed at improving functional recovery and quality of life in stroke survivors.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers were diagnosed with cerebrovascular disease, aged 18 years and above, both male and female.

1.1.2. Body mass index between 18.5-29.9 kg/m2 1.1.3. No history of falls in the 6 months prior to the study. 1.1.4. Able to follow instructions and consent to participate in the study. 1.1.5. Able to communicate with the researcher and provide information by themselves.

1.1.6. Able to walk continuously for at least 10 meters safely.

Exclusion Criteria:

* 1.2.1 Having undergone surgery to insert metal implants in the body, such as pacemakers, deep brain electrodes.

1.2.2 High blood pressure, uncontrolled heart disease, or having underlying diseases, such as osteoarthritis, arthritis, such as gout, rheumatoid arthritis, severe and affecting treatment.

1.2.3 Having a wound on the skull and abnormal sensation. 1.2.4 Having a history of injury or pain in the extremities. At a pain score of more than 5 out of a full score of 10, assessed by (Visual Analog Scale) 1.2.5 There is a condition of the inner ear that is disturbed, affecting balance, such as tinnitus.

1.2.6. There are unresolved vision and hearing problems. 1.3 Criteria for withdrawing volunteers from the research 1.3.1 If a volunteer experiences pain or discomfort during the test, the test will be stopped and the volunteer will be removed from the research immediately.

1.3.2 The volunteer requests to withdraw or is unwilling to continue the research.

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-04-20 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2025-01-30 (Actual)

PRIMARY OUTCOMES:
Change in Functional Mobility (TUG) | 4 week
  Balance control was measured using the Timed up and go test (TUGT). The tester measured the time it took the volunteers to stand up from a chair, walk straight ahead for 3 meters, turn around a cone, and walk back to sit in the chair at maximum speed and safety for 3 times. The average time taken by the volunteers in seconds was then calculated.
Change in Functional Mobility (10MWT) | 4 week
  Walking speed: The time taken to walk a distance of 10 meters (10-meter walk test: 10MWT) at normal and maximum speeds was measured. The tester measured the time taken for the 4 meters in the middle of the entire walkway. The test was repeated 3 times/speed and the average of each speed was calculated in meters/second. The movement was analyzed using a 2D (high-speed) motion analysis program.
Change in Functional Mobility ( 6MWT) | 4 week
  Functional endurance was measured using a 6-minute walk test (6MinWT) in which subjects walked as far as possible around a rectangular walkway. During the test, subjects were allowed to stand and rest without interrupting the test time. At the end of the test, the tester measured the distance covered by the subjects.
Change in Functional Mobility (FTSST) | 4 week
  Functional muscle strength test of the leg muscles using the Five times sit-to-stand test (FTSST) as quickly and safely as possible without using hands. The test was repeated 3 times and the average was calculated.
Change in Functional Mobility (BBS) | 4 week
  Berg Balance Scale (BBS), a healthcare provider gives a person 14 tasks, such as sitting to standing, standing unsupported, and reaching for objects, scoring their performance from 0 (unable to complete) to 4 (normal). The total score out of 56 indicates functional balance, with higher scores showing better balance and lower scores suggesting a greater risk of falling. The assessment takes about 15-20 minutes and requires simple equipment like a chair, stopwatch, and step stool
Change in Functional Mobility (Fugl-Meyer Assessment (FMA)) | 4 week
  The Fugl-Meyer Assessment (FMA) assesses motor function, sensation, balance, joint range of motion, and joint pain, typically in stroke patients, using a standardized 3-point scale (0=cannot perform, 1=performs partially, 2=performs fully) for each item. An examiner observes the patient's ability to complete tasks and assigns scores for the upper extremity motor (66 points), lower extremity motor (34 points), sensation (24 points), balance (14 points), and joint pain and range of motion (44 points each). The final score, a number out of a possible 226, indicates the level of recovery, with higher scores signifying better functional ability

SECONDARY OUTCOMES:
Change in Cognitive Function (Montreal Cognitive Assessment (MoCA)) | 4 week
  MoCA, an examiner guides a patient through 10 minutes of tasks testing various cognitive domains, including attention, executive function, memory, language, and orientation, by having them copy a cube, draw a clock, remember words, name animals, and identify similarities between objects. The test is scored out of 30 points, with a score of 26 or higher generally considered normal.
Change in Cognitive Function (Stroop test) | 4 week
  the Stroop Test, measure and compare the time and accuracy for reading color words, naming colors in a non-conflicting way, and naming the color of ink in which an incongruent color word is printed.Color-Word Task: This is the main task where participants name the ink color of a color word that is printed in an incongruent color (e.g., the word "RED" in blue ink. The administrator records the number of correct responses within a set time (e.g., 45 seconds) or the total time to complete a set number of items.
Change in Cognitive Function (Digit Span) | 4 week
  Digit Span, a participant is asked to repeat sequences of numbers either in the original order (forward) or in reverse order (backward), with the sequence length increasing for correct repetitions.

CONTACTS AND LOCATIONS:
Overall Officials: Chonticha Kaewjoho, PhD, Principal Investigator — University of Phayao
Locations (3):
- Thailand (3):
  - Mar Fah Luang university, Chiang Rai, Chiangrai
  - Narongsak Khamnon, Chiang Rai, Tha Sut
  - Chonticha Kaewjoho, Phayao